CLINICAL TRIAL: NCT06394674
Title: A Prospective, Randomized, Phase ll Clinical Trial of Single-agent Treatment With Different Doses of Sulfamethoxazole Furmonertinib in Patients With Advanced, Metastatic Lung Adenocarcinoma Who Have Progressed After First- or Second-line Treatment With EGFR-TKl Osimertinib
Brief Title: High-dose Furmonertinib in the Treatment in Patients With Advanced, Metastatic NSCLC With Progressed After First- or Second-line Treatment With Osimertinib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The General Hospital of Eastern Theater Command (Other); Shanghai Chest Hospital (Other); Fujian Provincial Hospital (Other); Shanghai Changzheng Hospital (Other); The First Affiliated Hospital of Bengbu Medical University (Other); The First People's Hospital of Changzhou (Other); Second Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2023-155
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: furmonertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Furmonertinib 160mg QD (Experimental): Furmonertinib (AST2818) 160mg QD. All patients enrolled into this group will receive furmonertinib 160mg daily.
  Interventions: Drug: Furmonertinib
- Group B: Furmonertinib 240mg QD (Experimental): Furmonertinib (AST2818) 240mg QD. All patients enrolled into this group will receive furmonertinib 240mg daily.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Drug: Furmonertinib
  Other Names: AST2818

SUMMARY:
This is a prospective, randomised, uncontrolled phase II clinical trial planned to include 84 subjects with metastatic lung adenocarcinoma that had progressed after first- or second-line treatment with Osmertinib, who were randomly assigned to trial group 1 and trial group 2, and were given Furmonertinib 160 mg and 240 mg once/day, orally, respectively, with efficacy evaluated every 6 weeks until disease progression, intolerable toxic side effects, or Subjects voluntarily withdrew informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic lung adenocarcinoma
* Progression of imaging-confirmed extracranial lesions after first- or second-line treatment with Osimertinib
* Previous genetic testing for a definite EGFR-sensitive mutation and imaging-confirmed extracranial lesion progression after first-line treatment with Osimertinib; or previous genetic testing for a definite T790M mutation and imaging-confirmed extracranial lesion progression after second-line treatment with Osimertinib.
* Pre-existing clinical benefit after treatment with Osimertinib, including CR, PR, SD (duration >6 months);
* Patients with at least 1 measurable lesion according to the criteria for evaluating the efficacy of solid tumors (RECIST 1.1)
* Normal functioning of major organs
* Pre-menopausal women of childbearing potential with a negative serum or urine pregnancy test within 7 days prior to the first dose of the drug
* Subjects volunteered and signed a written informed consent form.

Exclusion Criteria:

* Previous chemotherapy or immunotherapy
* Patients with non-lung adenocarcinoma, including squamous lung cancer or mixed histological types
* Progression of imaging-confirmed extracranial lesions after prior Osimertinib treatment with accessible treatment options after genetic testing
* Patients with symptomatic brain metastases, meningeal metastases or spinal cord compression
* Any unrecovered CTCAE > grade 1 toxicity reaction following prior Osimertinib treatment at the start of study drug therapy
* Other malignant tumors within 5 years or history of other malignant tumours; except effectively controlled basal cell carcinoma of the skin, carcinoma in situ of the uterine cervix, ductal carcinoma in situ of the breast, papillary carcinoma of the thyroid, superficial bladder tumors, etc.
* History of interstitial pneumonia with previous diagnosis
* Other circumstances that, in the judgement of the investigator, make them unsuitable for inclusion in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Analysis will occur when PFS maturity is observed at approximately 12 months from the first patient begin study treatment
  Objective Response Rate (ORR) (per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments) is defined as the number (%) of patients with response

SECONDARY OUTCOMES:
Progression-free survival (PFS) | The primary analysis of Progression-free survival (PFS) based on investigator assessment will occur when PFS maturity is observed at approximately 12 months after the first patient begin study treatment
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Progression-free survival (PFS) is defined as the time from beginning of study treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable Response Evaluation Criteria in Solid Tumors (RECIST) assessment.
Disease Control Rate (DCR) | Analysis will occur when PFS maturity is observed at approximately 12 months from the first patient begin study treatment
  Disease control rate (DCR) is defined as the percentage of subjects who have a best overall response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the Investigator.
Duration of Response (DoR) | Duration of Response analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 12 months from the first patient begin study treatment
  Duration of Response is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.

OTHER OUTCOMES:
Adverse Events | From the start of study drug to 30 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China